CLINICAL TRIAL: NCT03724266
Title: Effect of Using Nanochitosan Versus Calcium Hydroxide as Intracanal Medications on the Postoperative Pain and Apical Bone Healing
Brief Title: Effect of Using Nanochitosan Versus Calcium Hydroxide as Disinfectant on Pain and Apical Bone Healing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ahmed abdelmonam abd elmougoud, Phd student, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ahmed abdelmonam
Record Dates: First submitted 2018-10-24; First posted 2018-10-30 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Postoperative Pain; Healing
MeSH Terms: conditions — Pain, Postoperative | interventions — Chitosan; Calcium Hydroxide

STUDY DESIGN:
Intervention Model Description: postoperative pain after intervention
Who Masked: Participant, Outcomes Assessor
Masking Description: participants should be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chitosan (Experimental): chitosan as intracanal medication 0.2% in form of gel
  Interventions: Drug: Chitosan
- calcium hydroxide (Active Comparator): intracanal medication
  Interventions: Drug: Calcium Hydroxide

INTERVENTIONS:
Drug: Chitosan — chitosan will be used as intracanal medication
  Arms: chitosan
Drug: Calcium Hydroxide — intracanal medication
  Other Names: CaOH
  Arms: calcium hydroxide

SUMMARY:
Effect of Using Nanochitosan versus Calcium Hydroxide as Intracanal Medications on the Postoperative Pain and Apical Bone Healing

DETAILED DESCRIPTION:
PICO approach P (population): maxillary anterior teeth having necrotic pulp with symptomatic apical periodontitis with evidence of apical radiolucency (minimum size 2 mm x 2 mm).

I (intervention):0.2% nanochitosan as intracanal medication. C (control): calcium hydroxide paste intracanal medication.

O (outcome):

Primary outcome: postoperative pain at time interval 4, 12, 24, 48, 72 hours

Secondary outcome:

1. Postoperative pain, swelling, palpation, percussion and mobility at one week, 3, 6, 12 months
2. Number of analgesic tablets used at 4, 12, 24, 48, 72 hours and one week.
3. healing of apical periodontitis using CBCT at 3, 6, 12 months

ELIGIBILITY:
Inclusion criteria:

* Patients in good general health.
* Patient's age ranging between 20-40 years with no sex predilection.
* Maxillary anterior teeth with non-vital pulp and symptomatic apical periodontitis.
* Evidence of apical radiolucency (minimum size 2 mm x 2 mm).
* Patients' acceptance to participate in the study.

Exclusion criteria:

* Medically compromised patients with a severe systemic condition.
* Pregnant female patients.
* Patients who had taken any antibiotic or analgesics during the past 24 hours.
* Presence of a swelling because emergency management may include incision and drainage.
* Retreatment cases.
* Generalized periodontitis (calculus, deep pockets).
* Out of normal variations (open apex- severely curved canal- obstructed canal).

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
change in postoperative pain after intervention of chitosan: NRS | 4,12,24,27 hours
  pain assessed by numerical rating scale, pain will be assessed using a numerical rating scale (NRS) which is proven to be a simple, valid, and a reliable pain measurement tool. The NRS consists of a series of numbers from zero to 10 with the end-points representing the extremes of pain as "no pain" and "the worst possible pain". Patients will rank their pain level by making a mark on the number they thought it represented their pain. The pain intensity is assigned into four categorical scores: 1, no pain (score 0); 2, mild (scores 1-3); 3, moderate (scores 4-6); 4, severe (scores 7-10). Pain is evaluated preoperatively and postoperatively after the initial visit at 4, 12, 24, 48, 72 hours

SECONDARY OUTCOMES:
change in healing of apical periodontitis | 3,6,12 months
  linear measurment of apical radiolucency using cone beam computed tomography